CLINICAL TRIAL: NCT05874869
Title: Effectiveness of Dihydroartemisinin-piperaquine as Seasonal Malaria Chemoprophylaxis in Extended High Transmission Settings of Tanzania: an Open Cluster Randomized Clinical Trial.
Brief Title: Dihydroartemisinin-piperaquine for Seasonal Malaria Chemoprophylaxis in Tanzania
Acronym: SMC-DP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Mwaiswelo (Other Government)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); National Institute for Medical Research, Tanzania (Other Government); Hubert Kairuki Memorial University (Other)
Responsible Party: Sponsor-Investigator, Richard Mwaiswelo, Co-Principal Investigator, Tropical Pesticides Research Institute, Tanzania
Organization: Tropical Pesticides Research Institute, Tanzania (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MUHAS-REC-10-2019-062
Record Dates: First submitted 2023-05-04; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Malaria; Chemoprophylaxis; Underfive Children
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dihydroartemisinin-piperaquine (Active Comparator): Dihydroartemisinin-piperaquine will be administered to the intervention arm
  Interventions: Drug: Dihydroartemisinin-piperaquine
- Control (No Intervention): Individuals that will get malaria infection and present at the health facility with clinical signs and symptoms will be treated according to the Tanzania National Malaria Treatment guidelines using artemether-lumefantrine.

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine — The drug will be administered once a day for three consecutive days for three months (March, April, and May)
  Arms: Dihydroartemisinin-piperaquine

SUMMARY:
Background: Malaria prevalence has declined globally following the scale-up of the interventions, including insecticide-treated bed-net, indoor residual spraying, and prompt diagnosis and treatment with artemisinin-based combination therapy (ACT). Despite the gained success in the control, malaria has remained a major public health problem, particularly affecting children aged < 5 years in sub-Saharan Africa. Most of the malaria transmissions occur during the rainy season, a relatively short period. Intervention using antimalarial chemotherapy in children during the transmission season has been shown to prevent malaria-related morbidity and mortality. The World Health Organization has recommended seasonal malaria chemoprevention (SMC) using Sulphadoxine-pyrimethamine (SP) plus amodiaquine (AQ) in children aged 3-59 months in areas with highly seasonal malaria transmission. However, SP-AQ resistance is widespread in Tanzania. Therefore, this study will assess the effectiveness of Dihydroartemisinin-piperaquine (DHA-PQ) as SMC for the control of malaria among children in Tanzania.

Methods: Afebrile children aged 3-59 months from Nanyumbu and Masasi districts in the Mtwara region will be enrolled in an open cluster randomized clinical trial, administered monthly with a full course of DHA-PQ for three or four consecutive months during the high malaria transmission season of the three consecutive years. Three approaches of DHA-PQ SMC administration will be tested; a door-to-door approach using community health workers (CHWs), outreach visits using local health facilities clinicians/nurses, and village health posts using selected CHWs. Study participants will then be followed-up to evaluate the impact of the intervention on all-course of malaria morbidity and mortality; adverse events associated with the intervention; acceptability, adherence, coverage, and cost-effectiveness of the intervention; treatment-seeking behavior; and the risk of rebound after the withdrawal of the intervention. The primary outcome will be a prevalence of clinical malaria defined as the presence of fever (axillary temperature of 37.5 degrees Celsius) or a history of fever in the past 24 hours and the presence of P. falciparum asexual parasitemia at any density.

Findings: The findings will be disseminated through community meetings, seminars, local and international conferences, and publication in international journals.

Impact: The findings from this study will provide information on the effectiveness of DHA-PQ for seasonal prevention of malaria morbidity and mortality in children aged < 5 years in Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* being afebrile,
* willing to participate in the trial, and
* the ability to swallow oral medications.

Exclusion Criteria:

* a presence of an acute febrile illness or severe illness that impairs the ability to take oral medication
* HIV-positive child receiving cotrimoxazole prophylaxis,
* a child who has received a dose of antimalarial drug including dihydroartemisinin-piperaquine during the past month; and
* a history of allergy to DHA-PQ.

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13800 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of clinical malaria | 12 months
  Defined as the presence of any malaria-related signs/symptoms plus P. falciparum asexual parasitemia at any density. For it to be considered a clinical malaria there must be any signs or symptoms related to malaria infection and the presence of asexual P. falciparum parasites confirmed by mRDT or microscopy.

SECONDARY OUTCOMES:
Incidence of severe malaria | 12 months
  Defined according to the WHO criteria
Prevalence of malaria infection | 12 months
  Defined as the presence of asexual parasitemia. Individuals do not show any signs or symptoms related to malaria infection but they have asexual P. falciparum parasites confirmed by mRDT or microscopy.
Prevalence of anaemia | 12 months
  Prevalence of mild, moderate, or severe anaemia defined as an hemoglobin concentration of 11 g/dL, 8 g/dL, or 5 g/dL, respectively.
Prevalence of hospital admissions | 12 months
  Prevalence of individuals admitted to the health facility due to malaria infection during the SMC will be assessed. Hospital admission will be defined as a stay of at least 24 hours in hospital for treatment.
Prevalence of participants with any anthropometric indices. | 12 months
  The prevalence of children with anthropometric indices including wasting, stunting, or underweight as defined by WHO will be assessed before and after the three rounds of SMC and then compared.
Prevalence of household heads with positive health seeking behavior | 12 months
  Initiatives to seek treatment once feels sick. A questionnainne will be used to gather information from the household heads of the children involved in the study on what initiatives do they take when they or their children become sick.
Prevalence of molecular markers | 12 months
  Molecular markers of artemisinin and partner drugs resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Muhimbili University of Health and Allied Ssciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with individuals locally and globally following guidelines stipulated in the Data and Material Transfer Agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months
Access Criteria: Request to the PI

REFERENCES:
- [Derived] Mwaiswelo R, Ngasala B, Chaky F, Molteni F, Mohamed A, Lazaro S, Samwel B, Mmbando BP. Dihydroartemisinin-piperaquine effectiveness for seasonal malaria chemoprevention in settings with extended seasonal malaria transmission in Tanzania. Sci Rep. 2024 Jan 25;14(1):2143. doi: 10.1038/s41598-024-52706-z. PMID 38273019